CLINICAL TRIAL: NCT02979600
Title: Clinical and Biological Efficacy of Peanut Oral Immunotherapy
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-051
Record Dates: First submitted 2016-11-17; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Peanut Allergy
Keywords: Oral immunotherapy; Oral tolerance induction
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An oral tolerance induction (OTI) protocol is conducted at the allergy Unit of Saint Vincent Hospital of Lille (France) in standard care since 2006. This protocol consists in exposing patients to regularly increasing doses of allergen. This protocol induces an increase of the threshold reactive dose (the minimum dose of allergen that triggered a reactive reaction) and a decrease of the quantity of specific immunoglobulin E (sIgE) against peanut proteins. The protocol is ended when the patient reaches a threshold reactive dose of 2942mg of peanut proteins, corresponding to 14 peanuts of middle size, which is the maximum dose of peanut that can be found in standard product in France.

The investigators wish to study the evolution of the threshold reactive dose and of the sIgE of patients that have followed the OTI protocol. All the needed data are available in the medical records so the study will be conducted on retrospective data.

DETAILED DESCRIPTION:
Prevalence of food allergy is estimated at 3.5% in Europe. In particular, peanut allergy prevalence in France is between 0.3% and 0.75%, when it is 1% in the US, UK and Canada. Peanut allergy is a severe allergy, second behind tree nut allergy in the general population, with a risk of fatal reactions. The risk is especially high for young adults. It is also a long lasting condition with only 20% of natural healing that happened most of the time between 6 and 8y.o. These last years, the only proposed "treatment" was an elimination diet. However, it has been proved that it makes allergy severity worse, and sensitization and reactivity increase with time. Elimination diet can also lead to the apparition of avoidant/restrictive food intake disorders, and has a major impact on patient habits, causing patient quality of life to decrease.

In view of the risks and limits of an elimination diet and the low natural healing rate, a therapeutic alternative has been proposed with the development of peanut oral tolerance induction (OTI) protocols. As sublingual immunotherapies have low efficacies and as injection strategies have a high risk of severe allergic reactions, oral route is preferred. This strategy needs to ensure patients an increasing tolerance to the allergen, thus limiting the risks of anaphylactic shock at low doses, but also needs to ensure patient safety, with controlled risks of secondary reactions at home. It can be followed by young patients, its efficiency being increased. An OTI protocol is conducted at the allergy Unit of Saint Vincent Hospital of Lille (France) in standard care since 2006. It consists in daily giving small peanut doses to the patient, and to regularly increase those doses.

For this OTI protocol, an oral food challenge (OFC) is performed. This OFC allows the determination of the threshold reactive dose, i.e. the minimum dose of allergen that induces an allergic reaction. A safe dose of peanut is then determined that will be regularly eaten by the patient. Every 6 months, a new OFC is performed and thus a new threshold reactive dose is measured, and the dose to be eaten by the patient updated. The protocol is followed until the patient reaches an ideal dose of 2942mg of peanut protein, corresponding to 14 peanuts of middle size, which is the maximum dose of peanut that can be found in standard product in France. Of course, the protocol can also be ended if the patient decided so.

Although this protocol is performed in the allergy Unit of Saint Vincent Hospital, very few data are published on the subject. The aim of the study is to study the evolution of the threshold reactive dose and the evolution of the quantity of specific immunoglobulin E (sIgE) against peanut proteins (rAra h 1, rAra h 2 and rAra h 3) in patient that had followed the protocol.

The main objective of this study is to study the clinical efficiency of peanut OTI by measuring the evolution of the patient threshold reactive dose.

The secondary objective is to study the biological efficiency of peanut OTI by measuring the evolution of the dosage of sIgE against peanut proteins.

As the OFC and the IgE dosage are a standard part of the OTI protocol, all the data are obtained from the medical records. The study is retrospective and thus observational.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms when consuming peanuts, such as urticaria, asthma, angioedema, atopic dermatitis, dermo-respiratory syndrome or anaphylactic shock.
* Positive sIgE against r Ara h 2 dosage, i.e. r Ara h 2 >0.1
* Patients that had followed a peanut oral tolerance induction

Exclusion Criteria:

* No clinical symptoms or biological confirmation of a peanut allergy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Peanut allergic patients that have followed a peanut oral tolerance induction protocol at the allergy Unit of Saint Vincent Hospital of Lille (France) since 2005
Sampling Method: Non-Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the threshold reactive dose in milligrams | At inclusion, then every 6 months until a threshold reactive dose of 2942mg of peanut protein is reached (up to 7 years)
  During the OTI protocol, an oral food challenge is performed every 6 months. The dose that induce the first allergic reaction is reported. The protocol is followed until the patients get a threshold reactive dose of 2942mg of peanut protein, or until the patient decide to end it.

SECONDARY OUTCOMES:
Evolution of IgE dosages against Arah1, 2 and 3 | At inclusion, then every 6 months until a threshold reactive dose of 2942mg of peanut protein is reached (up to 7 years)
  Dosage of the specific IgE against peanut proteins, rAra h 1, rAra h 2 and rArah 3, that are performed every 6 months during the standard follow-up of the patients. The measures are done with ImmunoCAP laboratory system, Phadia, Uppsala, Sweden.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Seynave, MD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No